CLINICAL TRIAL: NCT07246889
Title: A Randomized, Double-blind, Multicenter Phase III Study to Evaluate the Efficacy and Safety of AHB-137 Injection in Participants With HBeAg-negative Chronic Hepatitis B Treated With Nucleos(t)Ide Analogues
Brief Title: Study of AHB-137 in Participants With Chronic Hepatitis B (CHB) Treated With Nucleos(t)Ide Analogues (NAs)(AUSHINE)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ausper Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-10-8006
Record Dates: First submitted 2025-08-12; First posted 2025-11-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AHB-137 (Experimental)
  Interventions: Drug: AHB-137; Drug: NA therapy
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: NA therapy

INTERVENTIONS:
Drug: AHB-137 — AHB-137 will be injected weekly by subcutaneous injection. There are 2 leading doses on day 4 and day 11.
  Arms: AHB-137
Drug: Placebo — Placebo will be injected weekly by subcutaneous injection.Two additional doses given on day 4 and day 11.
  Arms: Placebo
Drug: NA therapy — NA will be the background therapy. After stopping the AHB-137 or placebo injection, continue for another 12 weeks.

SUMMARY:
This study is a randomized, double-blind, multicenter phase 3 clinical trial to evaluate the efficacy and safety of AHB-137 injection in participants with HBeAg-negative CHB treated with NAs.

ELIGIBILITY:
Inclusion Criteria:

* Participants voluntarily participate in the study, and sign the Informed Consent Form (ICF) prior to screening, able to complete the study according to the protocol;
* At least 18 years of age at the time of signing the ICF;
* Body mass index met the requirements;
* HBeAg negative at screening;
* HBsAg or HBV DNA positive for at least 6 months;
* Meet relevant requirements for NAs treatment;
* 100 IU/mL < HBsAg ≤ 3000 IU/mL, HBV DNA < 100 IU/mL and liver function indicators meet the requirements;
* Effective contraception as required.

Exclusion Criteria:

* Clinically significant abnormalities other than a history of chronic HBV infection;
* Concomitant clinically significant other liver diseases;
* Previous/current manifestations of hepatic decompensation;
* Significant hepatic fibrosis or cirrhosis;
* Presence of protocol-specified laboratory abnormalities;
* History of malignancy or ongoing assessment of possible malignancy;
* Those allergic to AHB-137 or its components;
* Participants with recent major trauma or major surgery, or planning surgery;
* Those who are participating in another clinical trial, or have not undergone a protocol-specified washout period prior to this study;
* Prior/current use of prohibited medications;
* Inappropriate for participation in this trial as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with persistent HBsAg < limit of detection (LOD) and HBV DNA < lower limit of quantification (LLOQ) at the 24th week after all treatment for CHB was discontinued | 24 weeks after discontinuation of all CHB treatment

SECONDARY OUTCOMES:
Proportion of participants with persistent HBV DNA < LLOQ . | 24 weeks after discontinuation of all CHB treatment
Proportion of participants with persistent HBsAg < LOD and HBV DNA < LLOQ | Up to 60 weeks
Concentration of HBsAg, HBV DNA, HBV RNA, HBcrAg, HBsAb,HBeAg, HBeAb | Up to 60 weeks
Relapse rate after discontinuation of NAs therapy. | Up to 60 weeks
Safety: Number and percentage of participants with detectable anti-drug antibodies (ADA). | Up to 60 weeks
Safety: Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAE) and clinically significant examination results. | Up to 60 weeks
Plasma concentrations of AHB-137. | Up to 60 weeks
Sequencing of the Viral DNA and/or viral RNA analysis for detection of drug resistance in the target region of AHB-137 | Up to 60 weeks
Change from baseline in EuroQol Five-Dimension Five-Level Scale (EQ-5D-5L) scores in participants with HBV infection. | Up to 60 weeks
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Changes of the hepatitis B quality of life (HBQOL) instrument in participants compared with baseline. | Up to 60 weeks
  This scale has 31 items, including 7 dimensions: psychological status, expected anxiety, vitality, shame, infectivity, health vulnerability, and viral response. Each item is scored on a 5-point scale, with higher scores indicating a more severe impact of hepatitis B on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: AusperBio Clinical Trials, Study Director — AusperBio Investigational Site
Locations (28):
- China (28):
  - AusperBio Investigational Site, Hefei, Anhui
  - AusperBio Investigational Site, Beijing, Beijing Municipality
  - AusperBio Investigational Site, Chongqing, Chongqing Municipality
  - AusperBio Investigational Site, Fuzhou, Fujian
  - AusperBio Investigational Site, Xiamen, Fujian
  - AusperBio Investigational Site, Lanzhou, Gansu
  - AusperBio Investigational Site, Foshan, Guangdong
  - AusperBio Investigational Site, Guangzhou, Guangdong
  - AusperBio Investigational Site, Shenzhen, Guangdong
  - AusperBio Investigational Site, Liuchow, Guangxi
  - AusperBio Investigational Site, Nanning, Guangxi
  - AusperBio Investigational Site, Guiyang, Guizhou
  - AusperBio Investigational Site, Zunyi, Guizhou
  - AusperBio Investigational Site, Haikou, Hainan
  - AusperBio Investigational Site, Zhengzhou, Henan
  - AusperBio Investigational Site, Wuhan, Hubei
  - AusperBio Investigational Site, Changsha, Hunan
  - AusperBio Investigational Site, Nanjing, Jiangsu
  - AusperBio Investigational Site, Zhenjiang, Jiangsu
  - AusperBio Investigational Site, Nanchang, Jiangxi
  - AusperBio Investigational Site, Changchun, Jilin
  - AusperBio Investigational Site, Shenyang, Liaoning
  - AusperBio Investigational Site, Shanghai, Shanghai Municipality
  - AusperBio Investigational Site, Taiyuan, Shanxi
  - AusperBio Investigational Site, Xi’an, Shanxi
  - AusperBio Investigational Site, Chengdu, Sichuan
  - AusperBio Investigational Site, Kunming, Yunnan
  - AusperBio Investigational Site, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No